CLINICAL TRIAL: NCT07157579
Title: Study of Notch 1 Mutation in Chronic Lymphocytic Leukemia and Non-Hodgkin's Lymphoma Patient
Brief Title: Notch 1 Mutation in Chronic Lymphocytic Leukemia and Non-Hodgkin's Lymphoma Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hayam Gamal Ahmed, principle investigator, Sohag University
Other Study IDs: Soh-Med-25-8-2MD
Record Dates: First submitted 2025-08-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)- Non-Hodgins's Lymphoma (NHL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Detection of Notch1 mutation using real time pcr on bone marrow aspirate samples or peripheral blood samples. — Detection of Notch1 mutation using real time pcr on bone marrow aspirate samples or peripheral blood samples.

SUMMARY:
* Detection of Notch1 mutation in BM or peripheral blood of of patients with NHL
* Detection of Notch1 mutation in BM or peripheral blood of of patients with chronic lymphocytic leukemia .
* Comparison between expression of mutation in patient with CLL and NHL.

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukemia (CLL), is the most common leukemia in the western world. with a higher incidence in males (1.7:1),Current treatment strategies vary depending on disease burden, from active monitoring in asymptomatic patients, to targeted therapies in more advanced disease.

CLL is characterized by the clonal expansion of B cells with a characteristic immunophenotype (i.e., smIgweak, CD29+, CD23+, CD20weak) that slowly accumulate in peripheral blood, bone marrow, and lymphoid tissues mainly as a result of defects in the apoptosis machinery such as the overexpression of Bcl2 family anti-apoptotic proteins .

The clinical heterogeneity of CLL does reflect differences in the biology of the disease, particularly the IGHV mutational status and chromosomal alterations (i.e., del13q, del11q, trisomy 12 and del17p). Beside del17p/TP53 mutation which is the strongest CLL biomarker for response to therapy, other mutations (e.g., SF3B1, ATM, NOTCH1, BRIC3) have been reported to correlate with the outcome of the disease, but they are not actionable yet .

Non-Hodgins's lymphoma (NHL), the most common hematological malignancy worldwide, refers to a diverse class of B-cell and T-cell proliferations. NHL is differentiated from Hodgkin's lymphoma by different clinical characteristics and the absence of Reed-Sternberg cells and Cd15 and Cd30 staining on histology .

There are over 40 major subtypes, the most common types include indolent follicular lymphoma (FL) and aggressive diffuse large B-cell lymphoma (DLBCL). Each type is associated with unique driver genetic mutations (e.g., 14:18 translocation in FL, 11:14 translocation in Mantle Cell, 8:14 in Burkitts lymphoma ) and unique risk factors (Epstein-Barr Virus (EBV) for Burkitt's lymphoma, human T-cell lymphoma virus (HTLV-1) for T-cell lymphoma (de Leval et Jaffe,2020) The NOTCH gene was first named in studies of Drosophila melanogaster with notched wings in the 1910s, Homologs of NOTCH were then identified in multiple metazoans, and all these NOTCH homologs shared similar structures and signaling components.

ELIGIBILITY:
IncluInclusion criteria: approval to sign an informed written consent, patient with NHL and CLL .

Exclusion Criteria:

Refusal to sign an informed written consent, patient on chemotherapy sion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The studied individuals will be classified into 2 groups:
  Group (I): represent available number of CLL cases Group (II): represents available number of NHL cases
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
-Detection of Notch1 mutation in BM or peripheral blood of of patients with NHL and patients with chronic lymphocytic leukemia . - Comparison between expression of mutation in patient with CLL and NHL using real time pcr | baseline

IPD SHARING:
Plan to Share IPD: Undecided